CLINICAL TRIAL: NCT02681497
Title: Characteristics and Health Outcomes of Patients With Type 2 Diabetes Treated With Canagliflozin Added to Insulin Therapy in a Real-world Setting
Brief Title: Use of Canagliflozin in Conjunction With Insulin in a Real-world Setting
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Principal Investigator, Stewart Harris, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 2843175DIA4018_Harris
Record Dates: First submitted 2016-02-06; First posted 2016-02-12 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: canagliflozin; diabetes; SGLT2; real-world data
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a retrospective chart review study aiming to assess the characteristics and health outcomes of patients with type 2 diabetes treated with canagliflozin when used in addition to insulin therapy. Furthermore, the project aims to establish an EMR-based cohort of patients with type 2 diabetes mellitus (T2DM) treated with canagliflozin to allow for future longitudinal studies that investigate outcomes over a longer follow-up period, and whether canagliflozin (when used in addition to insulin therapy) has an impact on diabetes-related healthcare costs.

DETAILED DESCRIPTION:
This retrospective study will use data from an Electronic Medical Record (EMR)-based database (Web based Diabetes Records (Web DR) researchable database), which has been used to study patient's socioeconomic characteristics, treatment patterns and health outcomes of patients with diabetes. The Web DR de-identified researchable database contains integrated demographic, clinical and laboratory test result data of patients who received care from outpatient diabetes clinics in London, Ontario. The database includes more than 16,000 patients and their clinic visit information since 2000.

Adult individuals (age>=18) with type 2 diabetes receiving , registered in Web DR who have been treated with canagliflozin in conjunction with insulin therapy will be selected for this study. The baseline period will be 6 months to allow for more complete observation of comorbidities and medication use patterns.

The main objective of this project is to assess the characteristics and health outcomes of patients with type 2 diabetes treated with canagliflozin when used in addition to insulin therapy.

HbA1c, lipid, blood pressure, weight and other clinical indicators will be gathered from lab results during the baseline period closest to the date of canagliflozin prescription and follow up period (the last clinical value within the follow-up period and >=30 days after the start of the medication data will be selected.

The type of insulin used and dosages prescribed during the study follow-up period will be extracted from the database to examine the insulin dosage prescription pattern and understand the use of insulin with canagliflozin and its impact on clinical outcomes.

Furthermore, use of oral antihyperglycemic agents (metformin, sulfonylureas, thiazolidinedione, alpha-glucosidase inhibitors, meglitinides, Dipeptidyl peptidase-4 (DPP-4) inhibitors, bromocriptine) and injectable antihyperglycemic therapies (pramlintide, Glucagon-like peptide-1 (GLP-1) receptor agonists) will be measured during the 6 months baseline period and the follow-up period of 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 2DM >18 years of age, diabetes patients on insulin who initiated Canagliflozin due to a need of tighter glycemic control .

Exclusion Criteria:

* glomerular filtration rate (GFR)<45, pregnancy, type 1

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will use data from an EMR-based (Web DR) researchable database, which has been used to study patient's socioeconomic characteristics, treatment patterns and health outcomes of patients with diabetes. The Web DR de-identified researchable database contains integrated demographic, clinical and laboratory test result data of patients who received care from outpatient diabetes clinics in London, Ontario. The database includes more than 16,000 patients and their clinic visit information since 2000. Adult individuals (age>=18) with type 2 diabetes registered in Web DR who have been treated with canagliflozin in conjunction with insulin therapy will be selected for this study.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
change in HbA1c value | baseline and 6 months
  mean change in HbA1c value at 6 months from baseline

SECONDARY OUTCOMES:
change in weight (kg) | baseline and 6 months
  mean change in weight at 6 months from baseline will be assessed
change in blood pressure (both systolic and diastolic blood pressure) | baseline and 6 months
  mean change in blood pressure at 6 months from baseline will be assessed
change in glomerular filtration rate | baseline and 6 months
  mean change in glomerular filtration rate at 6 months from baseline will be assessed
change in Insulin dose | baseline and 6 months
  change in Insulin dose (units) at 6 months from baseline will be assessed
Evidence of diabetic ketoacidosis documented | within the first 6 months from baseline
  Number of evidence of diabetic ketoacidosis within the first 6 months from baseline will be assessed
Evidence of genital infections documented | within the first 6 months from baseline
  Evidence of genital infections within the first 6 months from baseline will be assessed
Evidence of hypoglycemia events documented | within the first 6 months from baseline
  Number of hypoglycemia events documented within the first 6 months will be assessed
Evidence of urinary tract infection (UTI) documented | within the first 6 months from baseline
  Evidence of urinary tract infection (UTI)s documented within the first 6 months will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Harris, MD,MPH,FCFP,FACPM, Principal Investigator — The Universtiy of Western Ontario
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No